CLINICAL TRIAL: NCT06779162
Title: ROTEM-based Optimization of Anticoagulation Regimens in Lung Transplantation
Acronym: ROAR-LT
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Jaromir Vajter, Director of Extracorporeal Life Support Center, University Hospital, Motol
Other Study IDs: ROAR-LT
Record Dates: First submitted 2025-01-04; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Anticoagulation; Lung Transplantation; Viscoelastic Properties; Unfractionated Heparin
Keywords: Anticoagulation; Lung Transplantation; Rotational Thromboelastometry; ROTEM; UFH; INTEM; HEPTEM; Clotting time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 65 subjects who underwent lung transplantation on ECMO: All 65 subjects received unfractionated heparin (UFH) for anticoagulation. Coagulation assessments were performed preoperatively (the nearest laboratory findings prior to lung transplantation), before ECMO cannulation (laboratory results after administering UFH and prior to ECMO cannulation), and throughout the ECMO run (after reperfusion of the first transplanted lung)

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is now a standard component of intraoperative support during lung transplantation, requiring anticoagulation management, typically with unfractionated heparin (UFH). While monitoring methods such as Activated Partial Thromboplastin Time (aPTT), Activated Partial Thromboplastin Time Ratio (aPTTr), Anti-Factor Xa Activity (anti-Xa), and Activated Clotting Time (ACT) are commonly used, a reliable bedside method remains elusive due to the unreliability of ACT at low UFH doses. This study evaluates the correlation among these monitoring methods and investigates the potential of the ROTEM Clotting Time INTEM/HEPTEM ratio (I/Hr) as a bedside alternative.

DETAILED DESCRIPTION:
Investigators conducted a comprehensive analysis of all lung transplant cases performed between December 8, 2022, and July 13, 2024, as part of the Prague Lung Transplant Program. This study was designed to assess the feasibility of using the ROTEM Clotting Time INTEM/HEPTEM ratio (I/Hr) as a reliable and practical bedside method for monitoring anticoagulation during lung transplantation procedures supported by extracorporeal membrane oxygenation (ECMO). Inclusion criteria focused on patients who underwent double lung transplantation, required intraoperative ECMO support, and had complete laboratory data available. Based on these parameters, investigators included 65 patients in our analysis.

All enrolled patients received unfractionated heparin (UFH) for anticoagulation management during their lung transplant procedures. Coagulation was closely monitored at three critical time points: preoperatively (using the most recent laboratory results prior to surgery), immediately before ECMO cannulation (following UFH administration but prior to initiating ECMO support), and during the ECMO run (after the reperfusion of the first transplanted lung). To ensure a comprehensive assessment, coagulation status was evaluated using a combination of methods: Activated Partial Thromboplastin Time (aPTT), Activated Partial Thromboplastin Time Ratio (aPTTr), Anti-Factor Xa Activity (anti-Xa), Activated Clotting Time (ACT), and the ROTEM Clotting Time INTEM/HEPTEM ratio (I/Hr).

In all cases, ECMO was initiated using a centrally cannulated approach. The drainage cannula was inserted through the right atrial appendage, while the return cannula was positioned in the ascending aorta. This configuration ensured optimal support and minimized complications during the intraoperative period. Extracorporeal circulation was facilitated using advanced devices, including Rotaflow I and Cardiohelp systems, both equipped with heparin-coated ECMO circuits to enhance biocompatibility and reduce clot formation.

Laboratory analyses of aPTT, aPTTr, and anti-Xa levels were performed in the institution's central laboratory, adhering to standardized methodologies to ensure accuracy and consistency. Bedside monitoring of ACT was carried out using the Werfen - HemoChron® system, which provided real-time feedback on clotting status during the procedure. Additionally, viscoelastic testing was performed to provide a detailed assessment of coagulation dynamics. This was primarily conducted using the Werfen - ROTEM® Sigma device, although the ROTEM® Delta device was employed in instances where the primary system was unavailable.

This study aims to establish the utility of the I/Hr as a novel, reliable, and bedside-appropriate method for anticoagulation monitoring during lung transplantation supported by ECMO. By comparing this approach to established monitoring methods, such as aPTT, anti-Xa, and ACT, investigators hope to identify a more effective strategy that aligns with the unique anticoagulation challenges posed by ECMO support. Investigator's findings could pave the way for standardized and improved anticoagulation protocols in lung transplant patients, ultimately enhancing clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* double lung transplant
* use of intraoperative ECMO
* complete laboratory findings

Exclusion Criteria:

* combined heart-lung transplantation
* single-lung transplantation
* lung transplantation without ECMO support
* intraoperative bleeding requiring discontinuation of anticoagulation therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 65 lung transplant cases between December 8, 2022, and July 13, 2024, conducted as part of the Prague Lung Transplant Program.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Can ROTEM be utilized as a bedside method for managing UFH anticoagulation dosing? | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  To evaluate the relationship between these monitoring methods: I/Hr, aPTT (s), aPTTr, anti-Xa (IU/mL), ACT (s), and to explore the potential of I/Hr as a bedside alternative to UFH monitoring. Correlations will be calculated between ROTEM parameter I/Hr and each of the following laboratory methods:
  I/Hr and aPTT, I/Hr and aPTTr, I/Hr and anti-Xa, I/Hr and ACT.
  This approach will assess the strength and consistency of the correlations, providing insights into the feasibility of using I/Hr as a reliable bedside alternative to standard laboratory methods.
Is there a correlation between I/Hr and aPTT? | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  As part of UFH anticoagulation therapy monitoring, I/Hr and aPTT (measured in seconds) will be assessed at all defined time points (every 60 minutes of ECMO run).
Is there a correlation between I/Hr and aPTTr? | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  As part of UFH anticoagulation therapy monitoring, I/Hr and aPTTr will be assessed at all defined time points (every 60 minutes of ECMO run).
Is there a correlation between I/Hr and anti-Xa? | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  As part of UFH anticoagulation therapy monitoring, I/Hr and anti-Xa (measured in IU/mL) will be assessed at all defined time points (every 60 minutes of ECMO run).
Is there a correlation between I/Hr and ACT? | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  As part of UFH anticoagulation therapy monitoring, I/Hr and ACT (measured in seconds) will be assessed at all defined time points (every 60 minutes of ECMO run).

SECONDARY OUTCOMES:
Correlation between the laboratory methods aPTT and aPTTr. | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  The relationship between aPTT (measured in seconds) and aPTTr will be assessed as part of UFH anticoagulation therapy monitoring at all defined time points (every 60 minutes of ECMO run).
Correlation between the laboratory methods aPTT and anti-Xa. | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  The relationship between aPTT (measured in seconds) and anti-Xa (measured in IU/ml) will be assessed as part of UFH anticoagulation therapy monitoring at all defined time points (every 60 minutes of ECMO run).
Correlation between the laboratory methods aPTT and ACT. | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  The relationship between aPTT (measured in seconds) and ACT (measured in seconds) will be assessed as part of UFH anticoagulation therapy monitoring at all defined time points (every 60 minutes of ECMO run).
Correlation between the laboratory methods aPTTr and anti-Xa. | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  The relationship between aPTTr and anti-Xa (measured IU/ml) will be assessed as part of UFH anticoagulation therapy monitoring at all defined time points (every 60 minutes of ECMO run).
Correlation between the laboratory methods aPTTr and ACT. | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  The relationship between aPTTr and ACT (measured in seconds) will be assessed as part of UFH anticoagulation therapy monitoring at all defined time points (every 60 minutes of ECMO run).
Correlation between the laboratory methods anti-Xa and ACT. | From the initiation of general anesthesia at the start of the lung transplant procedure until ECMO decannulation. Laboratory methods will be performed every 60 minutes from anesthesia initiation to ECMO cessation, lasting up to 6 hours.
  The relationship between anti-Xa (measured in IU/ml) and ACT (measured in seconds) will be assessed as part of UFH anticoagulation therapy monitoring at all defined time points (every 60 minutes of ECMO run).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital in Motol, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No